CLINICAL TRIAL: NCT06009640
Title: Integration of Intraoperative Neuromonitoring Into Laparoscopic Pelvic Nerve Decompression Surgery
Brief Title: Integration of Intraoperative Neuromonitoring Into Decompression Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Cansu Gundogdu, Specialist doctor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/514/220/8
Record Dates: First submitted 2023-08-11; First posted 2023-08-24 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Nerve Entrapments; Pelvic Pain
MeSH Terms: conditions — Nerve Compression Syndromes; Pelvic Pain | interventions — Intraoperative Neurophysiological Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative neurophysiological monitoring for decompression surgery (Experimental): we integrated intraoperative neuromonitoring system into laparoscopic lumbosacral plexus nerve decompression surgery and simultaneusly recorded nerve roots from lumbar 5 to sacral 4 during the operation. Diseases that cause pelvic nerve compression such as abnormal vascular conflict, aberrant priformis muscle, and endometriosis have settled in hard-to-reach deep areas of the pelvis. These areas can be accesed more easily with by laparoscopy, which provides better magnification and visualization. Sacral and sciatic nerves might be damaged when performing decompression surgery in these deep pelvic areas. Patients who gave informed consent and underwent surgical treatment for a proven diagnosis of lumbosacral plexus nerve entrapment were included in the study.
  Interventions: Device: Intraoperative neurophysiological monitoring with Nicolet Endeavor IOM Machine

INTERVENTIONS:
Device: Intraoperative neurophysiological monitoring with Nicolet Endeavor IOM Machine — Integration of intraoperative neurophysiological monitoring (IONM) into laparoscopic decompression surgery to protect pelvic nerves by continuously monitoring when they are at risk during surgery.
  Other Names: Nicolet Endeavor IOM Machine

SUMMARY:
To describe a novel technique by integrating the intraoperative neurophysiological monitoring (IONM) into laparoscopy to protect pelvic nerves by continuously monitoring when they are at risk during surgery.

DETAILED DESCRIPTION:
We integrated intraoperative neuromonitoring system into laparoscopic lumbosacral plexus nerve decompression surgery and simultaneusly recorded nerve roots from lumbar 5 to sacral 4 during the operation. Diseases that cause pelvic nerve compression such as abnormal vascular conflict, aberrant priformis muscle, and endometriosis have settled in hard-to-reach deep areas of the pelvis. Sacral and sciatic nerves might be damaged when performing decompression surgery in these deep pelvic areas. We described a novel technique by integrating the intraoperative neurophysiological monitoring (IONM) into laparoscopy to protect pelvic nerves by continuously monitoring when they are at risk during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms of chronic pelvic pain , dyspareunia, dysmenorrhea and severe, burning sharp pain on the lower extremity dermatomes, which had been present for at least one year were included.

Exclusion Criteria:

* Patients who underwent laparoscopic decompression surgery but did not give informed consent were not included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Pain score assessment with visual Analogic Scale (VAS) | 1 month
  Pain symptoms (Dysmenorrhea, dyspareunia, dyschezia, sciatic pain, chronic pelvic pain) were evaluated preoperatively , and re-evaluated at the postoperative first month.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gundogdu, M.D.Dr, Principal Investigator — Kartal Dr. Lutfi Kirdar City Hospital
Locations (1):
- Kartal Dr. Lutfi Kirdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No